CLINICAL TRIAL: NCT06686758
Title: A Trial Investigating the Efficacy and Safety of LC-Z300-01 on Proteinuria in Patients With Diabetic Kidney Disease
Brief Title: Efficacy and Safety of LC-Z300-01 on Proteinuria in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024SL109
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose LC-Z300-01 (Experimental): Sugar cane polysaccharide LC-Z300-01: 0.5g at a time, 2 times a day , 30 minutes before breakfast and dinner, Oral administration.
  Interventions: Dietary Supplement: Sugar cane polysaccharide
- high-dose LC-Z300-01 (Experimental): Sugar cane polysaccharide LC-Z300-01: 1.0g at a time, 2 times a day , 30 minutes before breakfast and dinner, Oral administration.
  Interventions: Dietary Supplement: Sugar cane polysaccharide
- control (Placebo Comparator): Identical placebo: 2 tablets, 2 times a day , 30 minutes before breakfast and dinner, Oral administration.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Sugar cane polysaccharide — Sugar cane polysaccharide
  Arms: high-dose LC-Z300-01; low-dose LC-Z300-01
Dietary Supplement: Control — placebo
  Arms: control

SUMMARY:
The purpose of this RCT is to investigate the efficacy and safety of Sugar cane polysaccharide LC-Z300-01 on proteinuria in participants with diabetic kidney disease (DKD).

DETAILED DESCRIPTION:
The incidence of diabetic nephropathy has shown a year-by-year increase, establishing it as the leading cause of uremia. Despite guideline-recommended therapies such as RAS inhibitors, patients with diabetic nephropathy continue to face elevated risks of disease progression, particularly when massive proteinuria persists. Early intervention through nephropathy management can effectively slow renal function deterioration, demonstrating substantial clinical value in mitigating uremia risk.

LC-Z300-01, a sugarcane-derived polysaccharide formulated as a dietary supplement, is being evaluated in this prospective, placebo-controlled, double-blind, randomized clinical trial. Sixty participants with confirmed diabetic nephropathy will be randomly allocated (1:1:1) to receive low-dose polysaccharide, high-dose polysaccharide, or placebo for 24 weeks of intervention and subsequent monitoring.

The predefined primary endpoint is the absolute change in uACR from baseline to week 24. Secondary endpoints encompass: (1) proportion of participants achieving ≥30% reduction in uACR versus baseline; (2) annualized eGFR decline rate; (3) HbA1c trajectory alterations; and (4) time-in-range (TIR) glycemic control metrics. Safety assessments will be conducted for all enrolled subjects receiving ≥1 administered dose.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years.
2. Clinically diagnosed type 2 diabetes mellitus with biopsy-proven or clinically confirmed diabetic kidney disease.
3. HbA1c ≤9% at screening.
4. Elevated albuminuria defined as either: uACR ≥30 mg/g on ≥2 occasions within 3 months or sustained proteinuria >300 mg/24-hour urine collection.
5. eGFR ≥60 mL/min/1.73 m² (CKD-EPI equation) at baseline.
6. Stable RAS blockade therapy meeting either: Maximum tolerated dose of ACE inhibitor/ARB for ≥4 weeks pre-screening or documented intolerance to ACEi/ARB (with nephrologist confirmation).
7. If using SGLT2 inhibitors and/or nonsteroidal mineralocorticoid receptor antagonists (ns-MRAs): stable regimen ≥4 weeks pre-enrollment or commitment to maintain dosing throughout study.
8. Capacity to provide written informed consent (self or via legally authorized representative).

Exclusion Criteria

1. Type 1 diabetes or secondary diabetes.
2. Acute metabolic complications within 6 months: diabetic ketoacidosis (DKA), hyperosmolar hyperglycemic state (HHS), severe hypoglycemia requiring hospitalization.
3. Various primary glomerular diseases, other secondary renal diseases (e.g. lupus nephritis, vasculitis renal damage, gouty nephropathy, obstructive nephropathy, chronic pyelonephritis, tumour-associated renal disease, polycystic kidney disease, etc.).
4. Patients with a history of autoimmune diseases that cause renal impairment (including but not limited to systemic lupus erythematosus, systemic small vessel vasculitis, rheumatoid arthritis, ankylosing spondylitis, dry syndrome, etc.).
5. patients who have received dialysis treatment for acute kidney injury within 6 months or who are expected to undergo dialysis during the study.
6. patients with a history of malignancy within 5 years.
7. participation in other clinical studies within 3 months.
8. Pregnant or lactating women.
9. hypersensitivity to any of the components of the interventions in this study.
10. alcohol or other drug abuse, and other conditions deemed by the investigator to be inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of change in patient uACR compared to baseline | 24 weeks
  Events based on uACR measure compared to baseline

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) slope | 24 weeks
  Based on eGFR ( by CKD-EPI formula ) slope
Change from baseline in HbA1c | 24 weeks
  Based on instrumental measurements of HbA1c
Change from baseline in glucose time in target range | 24 weeks
  Based on continuous glucose monitoring
The proportion of patients with uACR ≥30% lower than baseline | 24 weeks
  Based on UACR measure compared to baseline
Incidence of adverse reactions | Start of treatment until the end of the treatment for 12 weeks
  The proportion of patients with adverse reactions to the total population

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided